CLINICAL TRIAL: NCT02589977
Title: Myocardial Perfusion, Oxidative Metabolism, and Fibrosis in HFpEF
Acronym: HFpEF-PRoF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Marvin W. Kronenberg, M.D. (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Marvin W. Kronenberg, M.D., Professor of Medicine and Radiology, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 141686
Record Dates: First submitted 2015-08-24; First posted 2015-10-28 (Estimated); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-02

CONDITIONS: Heart Failure, Diastolic; Diastolic Heart Failure; Hypertension
Keywords: magnetic resonance imaging; positron-emission tomography; echocardiography; myocardial blood flow; energy metabolism
MeSH Terms: conditions — Heart Failure, Diastolic; Hypertension | interventions — regadenoson; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- normal participants (Other): No cardiovascular abnormalities or diabetes. Estimated glomerular filtration rate (eGFR) >60.
  Studies: Echocardiography for left ventricular function and LV diastolic performance; cardiac magnetic resonance (CMR) imaging using gadolinium for LV fibrosis and regadenoson for myocardial blood flow (MBF); positron-emission tomography (PET) using regadenoson for MBF and 11C-acetate for oxidative metabolism.
  Interventions: Drug: regadenoson
- hypertensive participants (Other): No history of coronary artery disease or diabetes. Estimated glomerular filtration rate (eGFR) >60.
  Studies: Echocardiography for left ventricular function and LV diastolic performance; cardiac magnetic resonance (CMR) imaging using gadolinium for LV fibrosis and regadenoson for myocardial blood flow (MBF); positron-emission tomography (PET) using regadenoson for MBF and 11C-acetate for oxidative metabolism.
  Interventions: Drug: regadenoson
- HFpEF patients (Other): No history of coronary artery disease or diabetes. Estimated glomerular filtration rate (eGFR) >60.
  Studies: Echocardiography for left ventricular function and LV diastolic performance; cardiac magnetic resonance (CMR) imaging using gadolinium for LV fibrosis and regadenoson for myocardial blood flow (MBF); positron-emission tomography (PET) using regadenoson for MBF and 11C-acetate for oxidative metabolism.
  Interventions: Drug: regadenoson

INTERVENTIONS:
Drug: regadenoson — evaluation of myocardial blood flow, interstitial fibrosis and oxidative metabolism in HFpEF, compared to hypertensive and normal participants
  Other Names: positron emission tomography; echocardiography; cardiac magnetic resonance imaging

SUMMARY:
Unlike heart failure with reduced ejection fraction (HFrEF) where several medicines and devices have been demonstrated to reduce mortality, no such therapies have been identified in HFpEF. This may be in part due to incomplete understanding of the underlying mechanisms of HFpEF.

Recently, impaired myocardial blood flow, reduced myocardial energy utilization, and increased myocardial fibrosis have been postulated to play important pathophysiologic roles in HFpEF. The investigators and others have demonstrated that HFrEF may be associated with altered myocardial energy utilization and "energy starvation." However, there are limited data regarding "energy starvation" in HFpEF and the relationships between myocardial blood flow, energy utilization, and fibrosis in HFpEF are largely unknown. Therefore, the purposes of this study are to use non-invasive cardiac imaging techniques to describe cardiac structure, function, blood flow, energetics, and fibrosis, and the relationships between these in order to better understand underlying mechanisms in HFpEF.

DETAILED DESCRIPTION:
The investigators hypothesize that HFpEF is associated with reductions in myocardial blood flow and energy utilization and increased myocardial fibrosis as compared to age and gender matched hypertensive and healthy controls. The investigators will test their hypotheses by comparing measurements of myocardial blood flow, energy utilization, and fibrosis between three subject groups (HFpEF vs hypertension vs healthy). Myocardial blood flow will be quantitated from nitrogen (N)13-Ammonia positron emission tomography (PET) and gadolinium enhanced cardiac magnetic resonance (CMR) imaging, both at rest and stress following coronary vasodilation with regadenoson. Myocardial energy utilization will be quantified with 11C-acetate PET imaging and myocardial fibrosis will be assessed with gadolinium enhanced CMR and alterations in myocardial T1. Echocardiography will be utilized to quantify cardiac diastolic function.

It is anticipated that the results of this proposed study will provide a foundation that will inform future studies aimed at identifying novel preventive or therapeutic agents in HFpEF.

ELIGIBILITY:
ALL

Inclusion Criteria:

* estimated glomerular filtration rate (eGFR) > 60 ml/min
* preserved left ventricular ejection fraction (>= 50%) on echocardiography

Exclusion Criteria:

* coronary artery disease
* diabetes mellitus
* contraindications to cardiac magnetic resonance imaging (CMR)
* weight >350 lbs
* inability to lie flat for imaging
* anemia
* contraindications to regadenoson or aminophylline

HEALTHY

Inclusion criteria:

* normal cardiac structure and function on echocardiography
* BP < 140/90

Exclusion criteria:

* known cardiovascular disease, cardiac risk factors or use of cardiac medications

HYPERTENSIVE

Inclusion criteria:

* history of BP >140/90
* 1 or more antihypertensive medications
* LV ejection fraction (LVEF) at least 50%
* current BP < 160/90

Exclusion criteria:

* known cardiovascular disease or risk factors aside from hypertension or use of cardiac medications

HFpEF

Inclusion criteria:

* physician-confirmed diagnosis of HF
* symptomatic HF
* LVEF at least 50%
* elevated LV filling pressure by catheterization, echocardiographic criteria or B-type-natriuretic peptide > 100
* current BP < 160/90

Exclusion criteria:

* prior history of LVEF below 50%
* acute decompensated HF
* moderate or greater valvular disease
* significant cardiac arrhythmias
* pericardial disease
* congenital heart disease
* primary pulmonary hypertension

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-11; Primary Completion 2020-01-21 (Actual); Study Completion 2020-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marvin W Kronenberg, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] Bell SP, Adkisson DW, Ooi H, Sawyer DB, Lawson MA, Kronenberg MW. Impairment of subendocardial perfusion reserve and oxidative metabolism in nonischemic dilated cardiomyopathy. J Card Fail. 2013 Dec;19(12):802-10. doi: 10.1016/j.cardfail.2013.10.010. Epub 2013 Oct 29. PMID 24331202
- [Result] Gupta DK, Shah AM, Castagno D, Takeuchi M, Loehr LR, Fox ER, Butler KR, Mosley TH, Kitzman DW, Solomon SD. Heart failure with preserved ejection fraction in African Americans: The ARIC (Atherosclerosis Risk In Communities) study. JACC Heart Fail. 2013 Apr;1(2):156-63. doi: 10.1016/j.jchf.2013.01.003. PMID 23671819

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Participants: No cardiovascular abnormalities or diabetes. Estimated glomerular filtration rate (eGFR) >60.
  Studies: Echocardiography for left ventricular function and LV diastolic performance; cardiac magnetic resonance (CMR) imaging using gadolinium for LV fibrosis and regadenoson for myocardial blood flow (MBF); positron-emission tomography (PET) using regadenoson for MBF and 11C-acetate for oxidative metabolism.
  regadenoson: evaluation of myocardial blood flow, interstitial fibrosis and oxidative metabolism in HFpEF, compared to hypertensive and normal participants
- Hypertensive Participants; HFpEF Patients: No history of coronary artery disease or diabetes. Estimated glomerular filtration rate (eGFR) >60.
  Studies: Echocardiography for left ventricular function and LV diastolic performance; cardiac magnetic resonance (CMR) imaging using gadolinium for LV fibrosis and regadenoson for myocardial blood flow (MBF); positron-emission tomography (PET) using regadenoson for MBF and 11C-acetate for oxidative metabolism.
  regadenoson: evaluation of myocardial blood flow, interstitial fibrosis and oxidative metabolism in HFpEF, compared to hypertensive and normal participants
Period: Overall Study
Arm/Group | Normal Participants | Hypertensive Participants | HFpEF Patients
Started | 23 | 20 | 12
Completed | 17 | 15 | 8
Not Completed | 6 | 5 | 4

BASELINE CHARACTERISTICS:
Population: These are the people who attended baseline visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Participants | Hypertensive Participants | HFpEF Patients | Total
Number analyzed (Participants) | 17 | 15 | 8 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 57 [54 to 62] | 58 [54 to 65] | 69 [62 to 73] | 58 [55 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 7 | 24
  Male | 5 | 10 | 1 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2
  White | 16 | 15 | 7 | 38
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 15 | 8 | 40
Hypertension [Count of Participants; unit: Participants] | 0 | 15 | 8 | 23
Diabetes [Count of Participants; unit: Participants] | 0 | 0 | 3 | 3
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 26.7 [22.6 to 28.7] | 30.1 [27.8 to 35.7] | 34.2 [29.9 to 37.8] | 29.7 [25.6 to 33.0]

OUTCOME MEASURES:

1. Primary Outcome: Coronary Flow Reserve
Description: Rest and regadenoson stress coronary flow reserve by ammonia PET. Coronary flow calculated at rest and again at stress with coronary flow reserve calculated as the ratio of stress to rest coronary flow.
Time Frame: Baseline study visit
Population: Incomplete data for 18 because of either inability to complete scan OR scan quality not adequate for analysis.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Normal Participants | Hypertensive Participants | HFpEF Patients
Number analyzed (Participants) | 10 | 6 | 6
ratio | 2.64 [2.34 to 2.85] | 2.65 [2.56 to 3.11] | 2.06 [1.96 to 2.26]

2. Secondary Outcome: Myocardial Perfusion Reserve by CMR in Each Study Group.
Description: Myocardial perfusion reserve by CMR.
Time Frame: Baseline study visit.
Population: Incomplete data for 10 because of either inability to complete scan OR scan quality not adequate for analysis.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Normal Participants | Hypertensive Participants | HFpEF Patients
Number analyzed (Participants) | 15 | 12 | 3
ratio | 2.19 [1.81 to 2.64] | 1.74 [1.44 to 2.59] | 1.29 [1.11 to 1.32]

3. Secondary Outcome: Extracellular Volume (ECV) by CMR in Each Study Group
Description: Extracellular volume (ECV) by CMR.
Time Frame: Baseline study visit
Population: Incomplete data for 9 because of either inability to complete scan OR scan quality not adequate for analysis.
Measure: Median (Inter-Quartile Range); unit: percent ECV
Arm/Group | Normal Participants | Hypertensive Participants | HFpEF Patients
Number analyzed (Participants) | 13 | 12 | 6
percent ECV | 31.9 [28.5 to 34.2] | 29.2 [27.4 to 33.1] | 30.9 [29.4 to 32.8]

4. Secondary Outcome: Oxidative Metabolism (Kmono/Rate Pressure Product) by PET in Each Study Group.
Description: Oxidative metabolism (Kmono/rate pressure product) by PET.
Time Frame: Baseline study visit
Population: Incomplete data for 4 because of either inability to complete scan OR scan quality not adequate for analysis.
Measure: Median (Inter-Quartile Range); unit: min-1/(beats/min x mmhg)
Arm/Group | Normal Participants | Hypertensive Participants | HFpEF Patients
Number analyzed (Participants) | 16 | 14 | 6
min-1/(beats/min x mmhg) | 0.12 [0.10 to 0.13] | 0.09 [0.07 to 0.11] | 0.09 [0.09 to 0.10]

5. Secondary Outcome: E/e' by Echo in Each Study Group.
Description: E/e' by echo. E is the transmitral peak velocity in early diastole. e' is the early diastolic tissue Doppler velocity average between the septal and lateral mitral annulus. E/e' is the ratio of these two values.
Time Frame: Baseline study visit
Population: We were able to collect data on all participants who completed the study.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Normal Participants | Hypertensive Participants | HFpEF Patients
Number analyzed (Participants) | 17 | 15 | 8
ratio | 7.2 [6.4 to 9.0] | 8.2 [7.2 to 9.4] | 13.0 [10.2 to 18.9]

ADVERSE EVENTS:
Time Frame: This is a cross sectional study. Subjects were followed for adverse events between screening/enrollment to one day following completion of the cardiac imaging study visit. Because this was not a longitudinal study with serial measurements of the end points the time between enrollment and cross sectional cardiac imaging study visit was variable for each subject in accordance with the study protocol. All subjects completed study procedures within thirteen months of enrollment.
Arm/Group | Normal Participants | Hypertensive Participants | HFpEF Patients
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/20 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/20 | 0/12
Other Adverse Events (participants affected / at risk) | 0/23 | 0/20 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/77/NCT02589977/Prot_SAP_000.pdf